CLINICAL TRIAL: NCT06440863
Title: The Effect of Changes in Body Mass Index After Total Knee and Hip Arthroplasty on Patient Functional Scores
Brief Title: Postoperative BMI Changes and Functional Outcomes in Knee and Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Mete Ozer, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y7MQG7gO
Record Dates: First submitted 2024-05-27; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Arthropathy; Obesity
Keywords: Total Hip Arthroplasty; Total Knee Arthroplasty; Weight Loss; Obesity; Body Mass Index
MeSH Terms: conditions — Joint Diseases; Obesity; Weight Loss | interventions — Arthroplasty, Replacement, Knee; Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Knee Arthroplasty (Active Comparator): Patients indicated for total knee arthroplasty.
  Interventions: Procedure: Total Knee Arthroplasty
- Total Hip Arthroplasty (Active Comparator): Patients indicated for total hip arthroplasty.
  Interventions: Procedure: Total Hip arthroplasty

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — Patients undergoing total knee arthroplasty
  Arms: Total Knee Arthroplasty
Procedure: Total Hip arthroplasty — Patients undergoing total hip arthroplasty
  Arms: Total Hip Arthroplasty

SUMMARY:
PURPOSE Obesity poses challenges to preoperative mobility and functional recovery for arthroplasty patients, yet postoperative weight loss remains elusive. This study aims to investigate postoperative weight changes and their impact on functional scores following knee and hip arthroplasty, exploring factors influencing these changes.

METHODS A total of 459 knee and hip arthroplasty cases with a 2-year follow-up were analyzed. BMI and Oxford scores were tracked, alongside factors including comorbidities, corticosteroid use, physiotherapy, and unilateral vs. bilateral surgery.

EXPECTED OUTCOMES Based on the study's design and the data available, we anticipate observing the impact of changes in patients' BMI on clinical scores as an independent variable. Additionally, we aim to elucidate the effects of comorbidities, corticosteroid use, physiatrist follow-up, and the type of surgical procedure on both BMI and clinical outcomes. Through this analysis, we expect to gain a comprehensive understanding of how these factors interplay to influence postoperative recovery and overall patient health.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent primary TKA and THA with a 2-year follow-up were included

Exclusion Criteria:

* Patients who underwent bariatric surgery before or after the surgery
* Incomplete 2-year follow-up
* Whom BMI or Oxford scores could not be accessed

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
BMI | 2 years
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters.
Oxford hip and knee scores | 2 years
  It is scored between 0 and 48. 48 is the best function.

CONTACTS AND LOCATIONS:
Overall Officials: Cumhur Deniz Davulcu, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University - Cerrahpasa, Cerrahpasa Faculty of Medicine, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Yes All demographic data, clinical scores, and BMI measurement results will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Woodruff MJ, Stone MH. Comparison of weight changes after total hip or knee arthroplasty. J Arthroplasty. 2001 Jan;16(1):22-4. doi: 10.1054/arth.2001.9826. PMID 11172266
- [Background] Riddle DL, Singh JA, Harmsen WS, Schleck CD, Lewallen DG. Clinically important body weight gain following knee arthroplasty: a five-year comparative cohort study. Arthritis Care Res (Hoboken). 2013 May;65(5):669-77. doi: 10.1002/acr.21880. PMID 23203539
- [Background] Inacio MC, Silverstein DK, Raman R, Macera CA, Nichols JF, Shaffer RA, Fithian D. Weight patterns before and after total joint arthroplasty and characteristics associated with weight change. Perm J. 2014 Winter;18(1):25-31. doi: 10.7812/TPP/13-082. PMID 24626069